CLINICAL TRIAL: NCT01555229
Title: Randomized, Single Blind Study Comparing the Effect of Intermittent Versus Continuous Subglottic Secretion Drainage on Tracheal Mucosa Damages in Intensive Care Patients Requiring Prolonged Mechanical Ventilation
Brief Title: Effect of Intermittent Versus Continuous Subglottic Secretion Drainage on Tracheal Mucosa Damages
Acronym: ASPIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrolment difficulties
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2010-A00912-37; CIC0203/124 (Other: RennesClinicalSearchCenter); LOC/09-05 (Other: Rennes University Hospital)
Record Dates: First submitted 2011-07-01; First posted 2012-03-15 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-04

CONDITIONS: Mechanical Ventilation Complication
Keywords: Secretion drainage; Ventilator-associated pneumonia; Tracheal fibroscopy
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent drainage (Experimental): Intermittent subglottic secretion drainage at -100 mmHg during 8 sec every 15 seconds.
  Interventions: Device: Intermittent subglottic secretion drainage
- Continuous drainage. (Active Comparator): Continuous subglottic secretion drainage at -20 mmHg.
  Interventions: Device: Continuous subglottic secretion drainage

INTERVENTIONS:
Device: Intermittent subglottic secretion drainage — Subglottic secretion drainage is performed using a specially designed endotracheal tube with a separate dorsal lumen that opens immediately above the endotracheal cuff.
  Arms: Intermittent drainage
Device: Continuous subglottic secretion drainage — Subglottic secretion drainage is performed using a specially designed endotracheal tube with a separate dorsal lumen that opens immediately above the endotracheal cuff.
  Arms: Continuous drainage.

SUMMARY:
Endotracheal tubes with subglottic secretion drainage (incorporating a suction port above the cuff) have been shown to reduce the incidence of ventilator-associated pneumonia. Subglottic secretion drainage can be either continuous or intermittent. However, concerns about the safety of continuous subglottic secretion drainage were raised in an experimental study in sheep, which found widespread injuries to tracheal mucosa and/or submucosa. Our objective is therefore to compare intermittent versus continuous subglottic secretion drainage on tracheal mucosa damages in patients requiring mechanical ventilation for an expected duration of more than 24 hours.

DETAILED DESCRIPTION:
Endotracheal tubes with subglottic secretion drainage (incorporating a suction port above the cuff) have been shown to reduce the incidence of ventilator-associated pneumonia. Subglottic secretion drainage can be either continuous or intermittent. However, concerns about the safety of continuous subglottic secretion drainage were raised in an experimental study in sheep, which found widespread injuries to tracheal mucosa and/or submucosa. Our objective is therefore to compare intermittent versus continuous subglottic secretion drainage on tracheal mucosa damages in patients requiring mechanical ventilation for an expected duration of more than 24 hours. Tracheal mucosa injuries will be assessed by tracheal fibroscopy. Secondary endpoints are the volume of daily secretions suctioned, the occurrence of difficulties or impossibilities of secretion drainage, and the occurrence of ventilator-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 years or more
* Patients hospitalized in intensive care unit
* Patients requiring endotracheal tube with an expected mechanical ventilation duration of more than 24 hours

Exclusion Criteria:

* Pregnant or breast-feeding women
* Previous known tracheal lesions
* Persons deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Tracheal mucosal damages assessed by tracheal fibroscopy. | the primary endpoint will be assessed just before extubation (variable duration depending on patient's status and cause of admission)
  * stage 0: no lesion
  * stage 1: erythema
  * stage 2 : oedema
  * stage 3 : ulceration
  * stage 4 : necrosis

SECONDARY OUTCOMES:
Volume of daily secretions | During intubation
Occurrence of difficulties or impossibilities of secretion drainage | During intubation
Occurrence of ventilator-associated pneumonia | During intubation

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Laviolle, MD, PhD, Study Chair — Rennes University Hospital; Philippe Seguin, MD, PhD, Principal Investigator — Rennes University Hospital
Locations (1):
- Service de Réanimation Chirurgicale, Hôpital de Pontchaillou, Rennes, France

REFERENCES:
- [Derived] Seguin P, Perrichet H, Pabic EL, Launey Y, Tiercin M, Corre R, Brinchault G, Laviolle B. Effect of Continuous versus Intermittent Subglottic Suctioning on Tracheal Mucosa by the Mallinckrodt TaperGuard Evac Oral Tracheal Tube in Intensive Care Unit Ventilated Patients: A Prospective Randomized Study. Indian J Crit Care Med. 2018 Jan;22(1):1-4. doi: 10.4103/ijccm.IJCCM_350_17. PMID 29422724